CLINICAL TRIAL: NCT00702455
Title: Novel Approaches to Weight Loss Maintenance
Brief Title: Keep It Off: A Weight Loss Maintenance Study
Acronym: KIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A06-025; 1R01CA128211 (NIH)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Weight Loss Maintenance
Keywords: Weight loss maintenance.; Interactive phone and mail-based intervention.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-Directed (Active Comparator)
  Interventions: Behavioral: Self-Directed (weight loss maintenance)
- Guided (Active Comparator)
  Interventions: Behavioral: Guided (weight loss maintenance)

INTERVENTIONS:
Behavioral: Self-Directed (weight loss maintenance) — Self- Directed participants will receive a core set of print materials describing key behaviors and skills necessary for successful weight loss maintenance and will review these materials with an intervention coach in two sessions.
  Arms: Self-Directed
Behavioral: Guided (weight loss maintenance) — Guided participants will receive 8 monthly check in calls and then bimonthly calls for the rest of the study. Guided participants are also asked to report their weight weekly, either via the Keep It Off website, email or voicemail. Those who experience weight gain will receive outreach calls to assist them in reversing their weight gain.
  Arms: Guided

SUMMARY:
The goal of this project is to test whether a phone and mail-based program designed to help people who have recently lost weight helps them keep the weight off over a 2 year period.

DETAILED DESCRIPTION:
Obesity is a major public health problem in the United States. Increases in obesity prevalence over the last four decades have been dramatic in all age and social groups, heightening concern about health risks for children, adolescents, and adults. Currently, over half of US adults are overweight and upward trends in prevalence show no sign of slowing. A continuation of current trends seems quite likely to lead to substantial increases in the number of people affected by obesity-related health conditions and in premature mortality. The primary treatment for obesity continues to be behavioral weight loss therapy, an approach that uses behavioral strategies (e.g., self-monitoring, stimulus control, problem-solving) to help participants adhere to dietary and physical activity recommendations. Significant progress has been made with respect to short term weight loss research over the past twenty years, with short term weight losses approximately doubling during this time period. Unfortunately, long term weight losses remain disappointing. The typical pattern is for maximum weight loss to occur at 6 months, with weight regain following. During the year following treatment, participants typically regain 30% to 50% of their initial weight loss. Follow-up beyond 1 year indicates a pattern of continued weight gain.

Though long term weight loss maintenance remains a critical challenge for obesity treatment, important information regarding successful weight loss maintenance (e.g., high levels of physical activity, self-weighing, maintenance of a low-fat, low-calorie diet) has been derived from the National Weight Control Registry led by Drs Wing and Hill. Treatment studies have incorporated such strategies to enhance maintenance; however, the most intensive treatment phase typically occurs during weight loss initiation with the maintenance phase occurring after treatment novelty has faded. Although increasing treatment duration improves weight loss, there is a point of diminishing returns as people eventually stop attending intervention sessions. An alternative strategy to provide the critical support necessary for weight loss maintenance may be to recruit people who have recently lost weight to a maintenance-focused intervention

We will recruit up to 400 adult men and women who have recently lost at least 10% of their body weight and randomize them to either a Self-Directed Intervention or a Guided Intervention . Self- Directed participants will receive a core set of print materials describing key behaviors and skills necessary for successful weight loss maintenance and will review these materials with an intervention coach during two phone sessions. Guided participants will take part in a set of ten core phone sessions addressing key factors relevant to weight maintenance (e.g., high levels of physical activity). After completing these sessions, Guided participants will receive 8 monthly check in calls and then bimonthly calls for the rest of the study. Guided participants are also asked to report their weight weekly, either via the Keep It Off website, email or voicemail. Those who experience weight gain will receive outreach calls to assist them in reversing their recent weight gain. They will also receive bi-monthly tailored feedback reports based on whether they are maintaining, losing or gaining weight. We hypothesize that those in the Guided arm of the study will regain less weight than those in the self-directed arm.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 19 and 70
* HealthPartners members for 11 out of the past 12 months
* Have lost at least 10% of body weight in the last 12 months

Exclusion Criteria:

* Lost weight via gastric by-pass surgery
* Modified Charlson scores >=3
* Nonskin cancer
* Congestive heart failure
* Coronary heart disease
* Psychotic illness
* Substance abuse
* Terminal illness
* Diagnosed eating disorder
* BMI<20.5 or >45

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Weight: Weight change in kilograms at 24 month follow-up. We hypothesize that Guided participants will regain less weight than the Self-Directed participants. | 24 months

SECONDARY OUTCOMES:
assessments of subgroup analysis of intervention effectiveness (e.g., BMI status, weight loss method, gender. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Sherwood, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Crain AL, Sherwood NE, Martinson BC, Jeffery RW. Mediators of Weight Loss Maintenance in the Keep It Off Trial. Ann Behav Med. 2018 Jan 5;52(1):9-18. doi: 10.1007/s12160-017-9917-x. PMID 28508330
- [Derived] Crane MM, Jeffery RW, Sherwood NE. Exploring Gender Differences in a Randomized Trial of Weight Loss Maintenance. Am J Mens Health. 2017 Mar;11(2):369-375. doi: 10.1177/1557988316681221. Epub 2016 Dec 5. PMID 27923968
- [Derived] Senso MM, Anderson CP, Crain AL, Sherwood NE, Martinson BC. Self-reported activity and accelerometry in 2 behavior-maintenance trials. Am J Health Behav. 2014 Mar;38(2):254-64. doi: 10.5993/AJHB.38.2.11. PMID 24629554